CLINICAL TRIAL: NCT05214625
Title: Questionnaire Study Concerning Artificial Intelligence and Its Application in (Gastrointestinal) Healthcare - Patients' and Physicians' Perspectives
Brief Title: Questionnaire Study Concerning Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Other Study IDs: METC 2020-2281
Record Dates: First submitted 2022-01-13; First posted 2022-01-31 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Gastro-Intestinal Disorders
Keywords: Artificial intelligence; Patients' perspective; Physicians' perspective; Questionnaire
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastroenterology patients: Patient receiving an endoscopic procedure because of regular care will be considered eligible for inclusion. Patients receive an endoscopic procedure in the context of the Dutch national screening program, because of gastrointestinal symptoms, or because of follow-up of previously diagnosed bowel diseases.
  Patients will be asked to complete a questionnaire concerning AI. No intervention will be administered.
  Interventions: Other: Questionnaire
- Gastroenterology physicians: GI physicians (both gastroenterologists and gastroenterology fellows), participating in a yearly gastroenterology and hepatology training day, will be asked for their participation in this study.
  Physician will be asked to complete a questionnaire concerning AI. No intervention will be administered.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire concerning artificial intelligence and its implementation in healthcare. GI patients and GI physicians will be provided with slightly different questionnaires.

SUMMARY:
This study aims to investigate the knowledge, experience, and opinion on AI among gastroenterology (GI) patients, gastroenterologists, and GI-fellows, particularly concerning implementation and application of AI (in assisting clinicians) in healthcare. The secondary aims are to investigate (dis)advantages of AI use in healthcare and the availability of technical facilities and infrastructures within endoscopy to implement and apply AI in Dutch hospitals.

DETAILED DESCRIPTION:
In recent years, important developments have been made in the field of artificial intelligence (AI). These developments have led to the large-scale application of AI in our everyday lives and AI-research within healthcare. A potentially promising application of AI lies in imaging analysis. For example, within gastroenterology this means the detection and classification of colorectal polyps and Barrett's neoplasia, disease severity scoring of inflammatory bowel diseases, and differentiating pancreatic cancer from chronic pancreatitis.

Despite the investments in AI-research, there is a lack in knowledge concerning patients' and physicians' perspectives on AI in healthcare. This prospective questionnaire study investigates these perspectives, obtaining data from both gastroenterology (GI) patients and GI-physicians within the Netherlands. The questionnaires focus on the knowledge, experience, and opinion of AI, particularly concerning the implementation of AI in (gastroenterology) healthcare. Furthermore, the current (endoscopic) infrastructure within Dutch hospitals will be investigated for its readnessy for AI.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal (GI) patients with an outpatient appointment in the gastroenterology department for an endoscopic procedure in the context of the Dutch national screening program, because of gastrointestinal symptoms, or because of follow-up of previously diagnosed bowel diseases (in one of the two participating hospitals);
* Gastroenterologists working in Dutch hospitals;
* Gastroenterology fellows working in Dutch hospitals;
* Minimal age of 18 years old.

Exclusion Criteria:

* No appropriate understanding of the Dutch language;
* Not willing to sign informed consent;
* Objection to participate in medical scientific research, reported in the medical file.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastroenterology patients who will have an outpatient appointment for an endoscopic procedure in the context of the national bowel cancer screening program, because of gastrointestinal symptoms, or because of follow-up of previously diagnosed bowel diseases, in one of two Dutch hospitals between April 2020 and September 2020.
  Gastroenterologists and gastroenterology fellows working in Dutch hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
The knowledge on AI investigated by means of a questionnaire | 6 months
  The knowledge on AI in healthcare among gastroenterology patients and physicians, investigated by means of a questionnaire.
The experience with AI investigated by means of a questionnaire | 6 months
  The experience with AI (in healthcare) among gastroenterology patients and physicians, investigated by means of a questionnaire.
The opinion on AI investigated by means of a questionnaire | 6 months
  The oninion on AI in healthcare among gastroenterology patients and physicians, investigated by means of a questionnaire.

SECONDARY OUTCOMES:
Willingness of physicians to use AI in (gastroenterology) healthcare | 6 months
  The willingness to apply AI in (gastroenterology) healthcare among gastroenterology physicians.
Willingness to apply AI in (gastroenterology) healthcare | 6 months
  The willingness of gastroenterology patients for their physicians to apply AI in (gastroenterology) healthcare.
Advantages and disadvantages of AI use in (gastroenterology) healthcare | 6 months
  Important advantages and disadvantages of AI use in (gastroenterology) healthcare among gastroenterology patients and physicians.
Potential domains within gastroenterology and hepatology for AI use | 6 months
  Potential domains within gastroenterology and hepatology for AI use indicated by GI physicians.
Mandatory infrastructure for AI use in healthcare | 6 months
  The availability of technical facilities and infrastructures within endoscopy to implement and apply AI in Dutch hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, Prof Dr MD, Principal Investigator — Maastricht Universitair Medisch Centrum
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study, including individual participant data, will be made available upon request. This data includes deidentified participant data. Additional documents that will be made available are the study protocol, the statistical analysis plan, the questionnaires, and the informed consent forms. Data will be available following publication with no end date. Requests should be methodologically sound proposals with the purpose to achieve aims in the approved proposal. Researchers who request the data should direct the proposal to q.vanderzander@maastrichtuniversity.nl to gain access. Data requestors will need to sign a data access agreement after approval of a proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following publication with no end date.
Access Criteria: Requests should be methodologically sound proposals with the purpose to achieve aims in the approved proposal. Data requestors will need to sign a data access agreement after approval of a proposal.

REFERENCES:
- [Background] Le Berre C, Sandborn WJ, Aridhi S, Devignes MD, Fournier L, Smail-Tabbone M, Danese S, Peyrin-Biroulet L. Application of Artificial Intelligence to Gastroenterology and Hepatology. Gastroenterology. 2020 Jan;158(1):76-94.e2. doi: 10.1053/j.gastro.2019.08.058. Epub 2019 Oct 5. PMID 31593701
- [Background] Shaban-Nejad A, Michalowski M, Buckeridge DL. Health intelligence: how artificial intelligence transforms population and personalized health. NPJ Digit Med. 2018 Oct 2;1:53. doi: 10.1038/s41746-018-0058-9. eCollection 2018. PMID 31304332
- [Background] Labovitz DL, Shafner L, Reyes Gil M, Virmani D, Hanina A. Using Artificial Intelligence to Reduce the Risk of Nonadherence in Patients on Anticoagulation Therapy. Stroke. 2017 May;48(5):1416-1419. doi: 10.1161/STROKEAHA.116.016281. Epub 2017 Apr 6. PMID 28386037
- [Background] Waymel Q, Badr S, Demondion X, Cotten A, Jacques T. Impact of the rise of artificial intelligence in radiology: What do radiologists think? Diagn Interv Imaging. 2019 Jun;100(6):327-336. doi: 10.1016/j.diii.2019.03.015. Epub 2019 May 6. PMID 31072803